CLINICAL TRIAL: NCT03283163
Title: Neurobiological and Psychological Benefits of Exercise in Chronic Pain and PTSD
Acronym: EXCPPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0704-W; 1k2 RX000704 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Chronic Musculoskeletal Pain; Posttraumatic Stress Disorder (PTSD); Mild or Moderate Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Lymphoma, Follicular | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: This study includes one group: Trauma-exposed participants suffering from both chronic musculoskeletal pain and varying degrees of PTSD severity. Those who meet diagnostic criteria for Chronic pain and have any symptoms of PTSD will be assigned to that group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic Pain//PTSD group (Experimental): This group of trauma-exposed participants with chronic musculoskeletal pain and varying degrees of PTSD severity will receive baseline and endpoint maximum load exercise testing which will inform their individualized exercise prescription (based on a progressive methodology) of aerobic exercise. Exercise training is aimed at meeting specific heart rate ranges over time (increasing up to 80% of maximum HRR between the midpoint and endpoint (6-12 weeks).
  Interventions: Behavioral: Exercise Testing and Training

INTERVENTIONS:
Behavioral: Exercise Testing and Training — The study group will perform a baseline maximum load exercise test which will inform the individualized exercise prescription for the participant. Based on a progressive methodology, the participant will engage in 12 weeks of exercise of their choice (walking, running, cycling or swimming) with the goal of working towards a maximum heart rate range of 80% between weeks 6 and 12 of the study.

SUMMARY:
The wars in Iraq and Afghanistan are creating a new generation of Veterans, including an increasing number of women Veterans, who present with comorbid PTSD and chronic pain conditions from recent deployment-related physical injuries and exposure to psychological trauma. Health behavior change has become increasingly important in treating these conditions and proactively preventing long-term negative health sequelae, in order to benefit these Veterans directly and reduce the growing challenges to the healthcare system. The proposed CDA-2 program of research will use an innovative translational research approach to study whether a chronic progressive -based exercise program will reduce chronic pain symptoms in patients with varying degrees of PTSD symptom severity and to elucidate and modify potential PTSD-related deficiencies in neurobiological and psychological responses to exercise to optimize the physical and psychological benefits of exercise for these individuals.

DETAILED DESCRIPTION:
Due to the COVID-19 pandemic, and after consultation with the appropriate research oversight, all study procedures are temporarily suspended as of 3/15/20.

This study will explicitly examine the effects of a 12-week progressive exercise training program on 1) the clinical symptoms of chronic pain and varying degrees of PTSD symptom severity, 2) anti-stress, anti-nociceptive neurohormones such as allopregnanolone + pregnanolone (ALLO +PA) in Veterans with trauma exposure, chronic pain and varying degrees of PTSD symptom severity. The revised study design includes a baseline cardiopulmonary exercise assessment (CPX) that will inform the exercise prescription for a 12-week "progressive exercise" training program, comprised of three 30-45 minute exercise sessions per week (walking or running, depending on the ability/capacity of the participant). Exercise sessions will be initially supervised by an exercise physiologist in the Clinical Studies Unit (CSU) at the VA Boston Healthcare System and then each participant will transition into the home. Intermittent telephone calls by the PI will provide additional motivational support and assistance with problem solving. Implementation of the prescribed exercise regimen will also be supported by the use of heart rate and actigraph monitors programmed for the participant to achieve their prescribed heart rate range (HRR). Finally, an "endpoint" maximum load exercise assessment will occur at week 13 in order to track measurable change for both psychological and neurobiological factors and to delineate their impact on pain indices and PTSD symptomatology. Both maximum load exercise tests will be performed in accordance with guidelines published by the American College of Cardiology. Measures of pain symptomatology will be implemented 30 minutes before and 30 minutes after exercise testing at baseline and endpoint. It is anticipated that differences in biological responses to aerobic and anaerobic exercise as illustrated by variability among the participants, with varying degrees of PTSD symptom severity, will predict differences in the psychological and pain-reducing benefits of aerobic and anaerobic exercise. Once identified, such factors could be augmented by modification of the exercise regimen in order to help enhance the ant-stress hormone levels for the pain/PTSD population and experience clinically significant reductions in their symptoms. In order to obtain sufficient power, the proposed recruitment is 23 participants. Data from this pilot work will be used to compute effect sizes in support of a future clinical trial incorporating individually prescribed exercise regimens and a motivationally based exercise behavior change intervention aimed at reducing pain and PTSD symptoms in our Veterans. Advanced education and training is sought by this CDA-2 award applicant in four broad areas: 1) psychophysiology of chronic pain and PTSD with a sub-focus on sex differences, 2) the neurobiology of chronic stress, PTSD, and pain, 3) exercise physiology and 4) the neuropsychology and neurobiology of traumatic brain injury (TBI). The combination of didactic and experiential training in these areas will serve the PI's long-term goal of becoming an independent scientist/practitioner in the VA focused on development of improved treatments for health conditions co-morbid with PTSD such as chronic pain and mild to moderate TBI. In the shorter-term, this CDA-2 will allow the PI to develop a more effective, motivationally based, exercise behavior change protocol that fosters long-term exercise compliance in patients with trauma-exposure, chronic pain and varying degrees of PTSD symptom severity.. This intervention will be used as an adjunct to cognitive interventions for these disorders to be further developed and studied via a larger VA, NIH, or DOD-funded grant for which the PI will apply in years 4-5 of the CDA2.

ELIGIBILITY:
Inclusion Criteria:

* Only Veteran and civilian participants in whom a physical examination, medical history, EKG, and baseline laboratory studies including urine toxicology screens indicate that maximum load exercise testing will be safe will be included in this study.
* Participants must be free of medications and other substances, (e.g., illicit drugs and alcohol) with effects that could hinder data interpretation for 2-6 weeks depending on the medication and frequency of use (which must be cleared by the PI's primary mentor).
* If on pain medications with short half-lives, must be off of them for 5 half-lives before testing, generally about 24 hours.
* Any participant with an ICD9 chronic pain diagnosis, with a musculoskeletal etiology, as confirmed by the study rehab medicine doctor, will be allowed for inclusion in the study.
* Also, any participant with a confirmed psychiatric diagnosis of PTSD

  * or have trauma exposure without a diagnosis of PTSD but some symptoms of PTSD, including subthreshold PTSD
  * other psychiatric conditions
* Individuals must meet for current chronic PTSD (>3 months ) as assessed by the CAPS 1-Month Diagnostic Version.

Exclusion Criteria:

* Veteran and civilian participants will be excluded from participation in the study if they have:

  * a life threatening or acute physical illness (e.g., cancer)
  * current schizophreniform illnesses or bipolar disorder
  * or active suicidal or homicidal ideation requiring clinical intervention.
* Women participants who are pregnant or are intending to become pregnant within the next six months will be excluded from participation.
* Individuals with current or past alcohol and/or substance dependence (less than three months from date of screening assessment) will be excluded.
* individuals without PTSD who have had greater than one major depressive episode or diagnosis of another serious psychiatric illness in their past, e.g.:

  * bipolar disorder or a schizophreniform disorder except for Psychosis not otherwise specified due to PTSD-related sensory hallucinations.
* Individuals seeking pain treatment such as surgical interventions or who have a neuropathic origin to their pain will also be excluded.
* Participants with chronic pain concerns that cannot tolerate exercising in a reclining bike and those who have had a clinical history of coronary artery disease or positive stress test
* Uncontrolled cardiac arrhythmia
* Moderate-to-severe aortic stenosis
* Severe arterial hypertension (systolic >200 mmHg, diastolic>110 mm Hg)
* More than first degree atrioventricular block also will be excluded from participation.
* Finally, participants who screen positive by answering all four items on the TBI assessment, will be excluded from participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica R. Scioli, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
This is a VA single site study. There are no plans to share the data outside of VA Boston Healthcare System, unless specifically requested and approved by authorized officials of VA, once the study has ended. Any data shared will be de-identified and subject to a data use agreement (DUA).
Supporting Information: CSR
Time Frame: Data will be available once the primary results are published. Data will be available per VA regulations.
Access Criteria: Upon request and completion of the DUA with approval by the VA IRB.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from 8/25/2014-3/20/2020 at the VA Boston Healthcare System, Women's Health Sciences Division (WHSD), National Center for PTSD (NCPTSD).
  Participants were receiving care in the VA Boston Healthcare System (VABHS) or recruited from the community. Inclusion criteria for the proposed study will permit the recruitment of women as well as men from all ethnic and racial backgrounds who are at least 18 years of age, and able to speak and understand English.
Groups:
- Chronic Pain/PTSD Group: This group of trauma-exposed participants with chronic musculoskeletal pain and varying degrees of PTSD severity will receive baseline and endpoint maximum load exercise testing which will inform their individualized exercise prescription (based on a progressive methodology) of aerobic exercise. Exercise training is aimed at meeting specific heart rate ranges over time (increasing up to 80% of maximum HRR between the midpoint and endpoint (6-12 weeks).
  Exercise Testing and Training: The study group will perform a baseline maximum load exercise test which will inform the individualized exercise prescription for the participant. Based on a progressive methodology, the participant will engage in 12 weeks of exercise of their choice (walking, running, cycling or swimming) with the goal of working towards a maximum heart rate range of 80% between weeks 6 and 12 of the study.
Period: Overall Study
Arm/Group | Chronic Pain/PTSD Group
Started (23 participants total were recruited into the study) | 23 (All participants were trauma exposed, met ICD9 or ICD10 definition for chronic musculoskeletal pain and had varying levels of PTSD symptom severity. A total of 23 eligible participants were enrolled into the study.)
Completed | 12
Not Completed | 11
Not completed — Lost to Follow-up | 1
Not completed — other life commitments | 6
Not completed — COVID-19 institution wide halting | 1
Not completed — Participants tested positive for illicit drugs on the day of the testing and/or training procedures | 2
Not completed — Participant found to not be forthcoming with screening/baseline assessments | 1

BASELINE CHARACTERISTICS:
Population: Characteristics: A cohort of 12 sedentary Veterans and civilians completed the full study and were trauma exposed and diagnosed with chronic pain and varying levels of PTSD severity.
Arm/Group | Chronic Pain//PTSD Group
Number analyzed (Participants) | 23
Age, Continuous [Median (Standard Deviation); unit: years] — The age was recorded from the SCID-5 assessment, taking the participant's date of birth and numerical age.
  years | 44.96 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants] — These data were collected from our demographic worksheet/questionnaire.
  Participants
    Female | 8
    Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 7
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants] — All data was collected in the Northeastern part of the United States at the VA Boston Healthcare System.
  Participants
    United States | 23
West Haven Yale Multidimensional Pain Inventory (WHYMPI) [Mean (Standard Deviation); unit: units on a scale] — The WHY-MPI has been demonstrated to be applicable across a variety of clinical pain conditions. Its brevity, validity/ reliability, self-report nature and ease of scoring make it ideal for both clinical and research purposes. The WHY-MPI is sensitive to change following rehabilitation. Please note only the interference subscale of the WHY-MPI will be administered. Scoring for each item is on a 0-6 scale; higher scores indicating greater symptom severity. Scoring includes summing up the scale items and dividing by the number of items to yield an average score of 0-6. Population: Two participants were found to test positive for illicit substances and one was found to not be forthcoming during assessments so they were excluded from the final analyses due to measurement of neurohormone data.
  units on a scale
    number analyzed (Participants) | 20
    (all) | 2.85 (1.67)
Posttraumatic Stress Disorder Checklist-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — The PCL is a 20-item self-report that assesses the extent to which an individual is bothered by each PTSD symptom during the past month using a 5-point Likert-type scale. The PCL-5 is undergoing validation, but the previous PCL based on DSM-IV had good sensitivity (.82) and specificity (.83). Score ranges 0-80, with higher scores representing higher severity (worse outcome). Population: Two participants were found to test positive for illicit substances and one was found to not be forthcoming with assessments and one participant had missing data so they were excluded from the final analyses due to measurement of neurohormone data. Some missing data for one participant was also observed.
  units on a scale
    number analyzed (Participants) | 19
    (all) | 26.21 (14.32)
Pain Catastrophizing Scale [Mean (Standard Deviation); unit: units on a scale] — All 13 items on the PCS were drawn from previous experimental and clinical research on catastrophic thinking in relation to pain experience. The factor structure of the PCS has been replicated in several investigations. Scores for each item are on a 0-4 scale with higher scores indicating greater symptom severity, the scores can range from 0-52 and a cutoff of 30 is indicative of a clinically relevant level of catastrophizing. Population: Two participants were found to test positive for illicit substances and one participant was found to not be forthcoming with assessments and were therefore excluded from the final analyses due to measurement of neurohormone data.
  units on a scale
    number analyzed (Participants) | 20
    (all) | 21.35 (14.28)
ALLO +PA at rest (Pre MAX-EX testing) [Mean (Standard Deviation); unit: pg/ml] — Allopregnanolone plus pregnanolone, together termed ALLO+PA, are anti-stress and antinociceptive GABAergic neuroactive steroids that are found to be lower in trauma exposed populations yet can be upregulated through intense sympathetic system activation such as acute, vigorous, exercise (i.e. maximum load exercise testing). Resting (five minutes before exercise testing) and peak levels (30 minutes after exercise testing) were collected through blood plasma collection. Population: While we had 23 participants at baseline; 2 participants tested positive for illicit substances, 1 participant was excluded due to not being forthcoming with assessments, 2 participants did not have chronic pain and 1 participant's assay results were not detectable at this time for which we are awaiting updated assay results. This resulted in a sample of n=17 for the analysis.
  pg/ml
    number analyzed (Participants) | 17
    (all) | 3532.53 (5042.86)
ALLO+PA at peak (30 minutes post MAX-EX testing) [Mean (Standard Deviation); unit: pg/ml] — Population: While we had 23 participants at baseline; 2 participants tested positive for illicit substances, 1 participant was excluded due to not being forthcoming with assessment, 2 participants did not have chronic pain and 1 participant's assay results were not detectable at this time, for which we are awaiting updated assay results. This resulted in a sample of n=17 for the analysis.
  pg/ml
    number analyzed (Participants) | 17
    (all) | 6175.29 (16670.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline: PTSD Checklist-5 (PCL-5)
Description: To be administered at: Endpoint Exercise Test Evaluation Session (week 13). The PCL is a 20-item self-report that assesses the extent to which an individual is bothered by each PTSD symptom during the past month using a 5-point Likert-type scale. The PCL-5 is undergoing validation, but the previous PCL based on DSM-IV had good sensitivity (.82) and specificity (.83). Scoring for each item is on a 0-4 scale with higher scores indicating higher symptom severity. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Initial research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD across samples. However, additional research is needed. Evidence for the PCL for DSM-IV suggests that a 5-10 point change represents reliable change (i.e., change not due to chance) and a 10-20 point change represents clinically significant change.
Time Frame: Baseline and endpoint (at 13 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain//PTSD Group
Number analyzed (Participants) | 11
units on a scale | 15.64 (11.34)
Statistical Analysis 1: Comparison: Chronic Pain//PTSD Group; paired samples t-test to compare PTSD severity from baseline to endpoint (week 13); Test type: Other; p = .040, t-test, 2 sided

2. Primary Outcome: Change From Baseline: West Haven-Yale Multidimensional Pain Inventory- Interference Subscale (WHY-MPI)
Description: The WHY-MPI has been demonstrated to be applicable across a variety of clinical pain conditions. Its brevity, validity/ reliability, self-report nature and ease of scoring make it ideal for both clinical and research purposes. The WHY-MPI is sensitive to change following rehabilitation. Please note only the interference subscale of the WHY-MPI will be administered in this study. Scoring for each item is on a 0-6 scale; higher scores indicating greater symptom severity. Scoring for this measure includes summing up the items of the scale and dividing by the number of items for that scale to yield an average score of 0-6.
Time Frame: Baseline and endpoint (at 13 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain//PTSD Group
Number analyzed (Participants) | 12
units on a scale | 2.56 (1.63)
Statistical Analysis 1: Comparison: Chronic Pain//PTSD Group; paired samples t-test to compare degree of pain-related interference from baseline to endpoint (week 13); Test type: Other; p = .69, t-test, 2 sided

3. Primary Outcome: Change From Baseline: Pain Catastrophizing Scale
Description: The PCS-R is a 13-item measure of which items were drawn from previous experimental and clinical research on catastrophic thinking in relation to pain experience Factor analyses of the PCS have shown that catastrophizing can be viewed as a multidimensional construct comprising elements of rumination ("I can't stop thinking about how much it hurts"), magnification ("I worry that something serious may happen"), and helplessness ("There is nothing I can do to reduce the intensity of the pain"). The factor structure of the PCS has been replicated in several investigations. Scores for each item are on a 0-4 scale with higher scores indicating greater symptom severity, the scores can range from 0-52 and a cutoff of 30 is indicative of a clinically relevant level of catastrophizing.
Time Frame: endpoint (at 13 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain//PTSD Group
Number analyzed (Participants) | 12
units on a scale | 13.92 (12.06)
Statistical Analysis 1: Comparison: Chronic Pain//PTSD Group; paired samples t-test to compare severity of pain catastrophizing from baseline to endpoint (week 13); Test type: Other; p = .098, t-test, 2 sided

4. Secondary Outcome: ALLO+PA Resting (Pre-MAX-EX Testing) Post 12 Weeks of MAX-EX Testing
Description: ALLO+PA are anti-stress and antinociceptive neurosteroids that were measured in plasma at rest and peak (before and after a baseline and endpoint cardiopulmonary exercise test). Higher scores reflect greater levels of the anti-stress, antinociceptive neurohormone, indicating a better outcome.
Time Frame: 13 week endpoint Cardiopulmonary Exercise Test Session (MAX-EX)
Population: Trauma exposed participants with chronic musculoskeletal pain and varying degrees of PTSD symptom severity.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Chronic Pain//PTSD Group
Number analyzed (Participants) | 12
pg/ml | 5855.33 (6542.71)
Statistical Analysis 1: Comparison: Chronic Pain//PTSD Group; paired samples t-tests were conducted for comparison of resting ALLO+PA levels from baseline to endpoint (week 13); Test type: Other; p = .194, t-test, 2 sided

5. Secondary Outcome: ALLO+PA Peak (Pre-MAX-EX Testing) Post 12 Weeks of MAX-EX Testing
Description: as for outcome 4
Time Frame: 13 week endpoint Cardiopulmonary Exercise Test Session (MAX-EX)
Population: Trauma exposed participants with chronic musculoskeletal pain and varying degrees of PTSD symptom severity.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Chronic Pain//PTSD Group
Number analyzed (Participants) | 12
pg/ml | 4062.50 (5971.54)
Statistical Analysis 1: Comparison: Chronic Pain//PTSD Group; paired samples t-tests were conducted for comparison of peak ALLO+PA levels (30 minutes post MAXEX) from baseline to endpoint (week 13); Test type: Other — paired samples t-test; p = .343, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entire period of active recruitment for each participant (i.e., from the date of study entry through the follow-up, yielding a total of 8 months.
Arm/Group | Chronic Pain/PTSD Group
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Pain/PTSD Group (N=23)
1mm ST segment Depression on ECG during Exercise Test (Cardiac disorders) | 1 (1) — Conservatively, we stopped test for immediate evaluation by study cardiologist and subsequent referral to clinical cardiologist for follow-up. Per protocol (ACSM guidelines), >2mm ST segment depression is a criterion to stop the test.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Pain/PTSD Group (N=23)
Leg pain during exercise training phase of the study based on prior injury (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant experienced an increase in leg pain stemming from a prior injury years ago that flared up after an exercise training session. The participant was discontinued from study for follow-up to confirm no new injury occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03283163/Prot_SAP_000.pdf